CLINICAL TRIAL: NCT04465799
Title: "Efficacy of ENTREN-F Program: A Psycho-family and Multidisciplinary Intervention for Children From 8 to 12 Years Old With Childhood Obesity: A Controlled and Randomized Clinical Trial"
Brief Title: Efficacy of ENTREN-F Program: A Psycho-family Intervention in Childhood Obesity
Acronym: ENTREN-OB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Fondation de France (Other); NAOS Institute of Life Science (Industry); Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Ana Rosa Sepúlveda García, Principal Investigator. Senior Lecturer and Researcher., Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSI201679471R Science Ministry; Ref00099489. 2019-ES-000-6711. (Other Grant/Funding Number: Alcampo Foundation for Youth (Foundation of France))
Record Dates: First submitted 2020-04-14; First posted 2020-07-10 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; psycho-family intervention; controlled and randomized clinical trial; emotional regulation
MeSH Terms: conditions — Pediatric Obesity; Emotional Regulation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: ENTREN is based on a exhaustive previous literature review. It uses a cognitive-behavioural perspective, has a duration of 6 months and includes a module for children treatment centred on emotional regulation. Some contents from "LEARN Program for Weight Management" were adapted to childhood stages for the ENTREN programme, which includes five main dimensions: lifestyle, physical activity, health attitudes, social relationships, and nutrition. Spanish health guidelines from the Health Ministry, aimed to promote healthy eating habits and physical activity, were also taken into account. Motivational interviewing techniques have also been integrated into the sessions to promote children's and families' commitment to their health. Specifically, family content has been developed to adapt parental democratic educational style and improve communication with their children. A previous pilot study of ENTREN programme was conducted to describe its feasibility and acceptability in Primary Care.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ENTREN Programme (Experimental): This intervention consists in a total of 12 biweekly sessions: 9 sessions of 2-hr only for children, with a further three 3-hr sessions attended by both families and children together: nutrition, physical activity sessions, and a closing event session. Children content was developed based a cognitive-behavioural perspective, and included motivational interviewing tools. The aim of the children's programme is, to promote healthy eating habits, problem awareness, motivation to change unhealthy behaviours, health commitment, emotional regulation, social skills and self-esteem. One 2-hr session at 6, 12 and 18-month follow-up was provided to refresh skills, their physical activity, and nutritional behaviours.
  Interventions: Behavioral: ENTREN
- ENTREN-F Programme (Experimental): ENTREN-F has the same children's intervention than ENTREN. It has extra 6 2-hr sessions to work on family environment and communication, plus three 2-hr sessions attended by both families and children together. One 2-hr session at 6, 12 and 18-month follow-up was provided to refresh skills, their physical activity, and nutritional behaviours.
  Interventions: Behavioral: ENTREN-F
- Control group (Other): The intervention of this group consists in usual treatment in Primary Care provided by Endocrinology Services. 3 monthly face-to-face consultations and continuous online monitoring are provided to these families, oriented to promote healthy habits of nutrition and physical activity for 6 months. It works from an exclusively behavioural perspective. A token economy is used with the families as a system of contingency management based on the systematic reinforcement of target behaviour.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: ENTREN — ENTREN intervention for children (cognitive-behavioral perspective + motivational interview)
  Arms: ENTREN Programme
Behavioral: ENTREN-F — ENTREN intervention for children + family intervention.
  Arms: ENTREN-F Programme
Behavioral: Control group — Behavioral modification of habits
  Arms: Control group

SUMMARY:
ENTREN-F Programme describes a novel structured psychosocial family-based intervention from Primary Care using a train trip metaphor aimed at improving healthy lifestyles for the whole family. It is oriented to children aged 8-12 years old who have overweight or obesity. The ENTREN-F intervention lasts 6 months and consists in 12 biweekly 2-h2 sessions in group, following a multidisciplinary perspective.

The main aim is to examine the efficacy of the intervention program 'ENTREN-F' (intervention for children plus family intervention) on anthropometrics, behaviour, psychological and family factors, from a multidisciplinary perspective, compared with another group participating in the same program 'ENTREN' (intervention for children without family intervention) and with a control group (usual treatment) among Spanish children with overweight and obesity. Finally, (2) the second aim was to evaluate whether the changes were maintained 6, 12 and 18 months after the end of the intervention.

Hypothesis The specific hypotheses of the present study were as follows: (a) There will be significant differences in the adherence to treatment, being higher in the ENTREN-F group (b) There will be improvements in clinical outcomes regarding the anthropometric variables of the child, the level of physical activity, psychological distress, and eating disorder of the child, after both interventions (ENTREN and ENTREN-F programme), in comparison to control group (d) There will be only improvements in clinical outcomes regarding in the family's healthy life-style, psychological distress of the parents, and the family environment, after the intervention of the ENTREN-F programme. (e) The significant changes produced will remain stable at the 6,12 and 18-month follow-up in the ENTREN-F group.

DETAILED DESCRIPTION:
Sample: The sample will be made up of 240 children of 8-12 years old (IMC>P90). The dropout rate is expected to be 20%. The majority of the participants will be recruited through Primary Health Care Services, in collaboration with Paediatrics Area. A small percentage of the sample contacted the program after receiving information from their school or advertising posters. After assessment, they are assigned randomly to one of the three conditions.

For Patient Registries:

* Spanish Ministry of Economy, Industry and Competitiveness provides an annual quality assurance for monitoring and auditing all financial projects (4-yr). This plan addresses data validation and registry procedures.
* A review of databases is regularly scheduled.
* Sample size assessment has been verified, specifying the number of participants necessary to demonstrate an effect (size effect; N=240). Regarding the sample size, assuming a two-tailed test α = .05 and a power (1 - β) of .80, estimating a 23% difference in the prevalence rates of childhood obesity, and applying a correction of according to the guidelines of Browner, Newman, Cummings and Hulley (2007) to anticipate a possible sample loss of approximately 20%, based on the study by Robertson (2008), a sample size of 80 children per group has been estimated (n = 240). Therefore, it is expected to collect substantial changes with an N = 60 in each of the groups at the end of the 12-month follow-up.
* A preliminary statistical analysis plan has been described with the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan. A preliminary plan for missing data has also taken into account and missing values will be taken into account in analyses. An expert methodologist collaborates in the Project and advises us in this field of work.
* Standard operating procedures to address registration operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, adverse event reporting, and change management. All members of the Project has received a specific training by A.R.S.
* A data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used and normal ranges if relevant. This document is provided to the principal members of the team.

Assessment: The clinical evaluation consists in an interview where socio-demographic and family clinical variables are evaluated, the semi-structured child diagnostic interview is carried out (K-SADS-PL) based on Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and a battery of questionnaires are administered to the child and both parents. Assessment are carried out over time (T0 baseline vs. T1 post/6-month vs.T2, T3 and T4, 6, 12 and 18-month follow-up, respectively).

Multidisciplinary team: Most of the sessions of the psycho-family sessions workshop group and the psychological workshop group with children are conducted by psychologists, with at least Clinical Psych MSc, some of them also doing Clinical Psych PhD. All therapists have received specific training prior to the protocol and work from Motivational Interview perspective. The team also has a nutritionist, psychiatrist and an expert in physical activity, training in Motivational Interview. Finally, paediatricians and nurses from the health centres in the area collaborate actively in the Project. Meetings for feedback about the progress of the project and annual specialist seminars are organized. The results and progress are also shared in Paediatrics and Psychology conferences. A multidisciplinary project from Primary Care, combining the joint effort of different professionals that allows a rapid and effective overweight patient care protocol to be developed. Interest has grown in the Project by international PhD students and Postgraduate students as evidenced in their project collaboration and consequent training.

Relevance of the study: Overall, this project will represent a significant contribution to the scientific understanding of this field as well as a significant savings in economic costs derived from this illness. It is expected to have an important clinical impact in the Madrid region, providing assistance to 240 families in the hospital. This is a pioneer research project that examines the efficacy of the new program of psychosocial family-based intervention for childhood overweight and obesity within Primary Care. The innovation and creativity of the ENTREN program for children highlights the broad content in emotional self-regulation, which has two aims: it helps to overcome the emotional difficulties (frustration, anxiety, impatience) and modify their eating habits, in turn, it could help to reduce the onset of unhealthy eating patterns or their prevalence (binge eating, emotional eating, picking). In addition, it highlights the inclusion of the family as a key factor in the change and implement of healthy lifestyles in children with overweight/obesity. The programme ENTREN-F (pilot study results) has been awarded by the Ministry of Health and Consumer Affairs, Strategy for Nutrition, Physical Activity and Prevention of Obesity (NAOS annual Award) in December 2017.

Ethical approval: The study received ethical approval by the Child and Adolescent Hospital Niño Jesús (Ref. R-0058/16), Central Committee of Research, Primary Care Commission (Ref. 32/17; 13.12.17) and Autonomous University Ethics approval (CEI-76-1394).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 8-12 years
2. BMI > Percentile 90
3. Presenter of physical and cognitive development according to sex and age
4. Good understanding of Spanish orally and in writing.
5. Do not present any difficulty that prevents the performance of autonomous physical activities

Exclusion Criteria:

1. standing obesity caused by a genetic syndrome
2. the child or none of their primary caregivers do not have adequate command of oral or written Spanish

a) Intellectual disability b) dieting supervised by an endocrine specialist at the time of the evaluation c) To suffer a serious psychological or medical disorder that requires immediate intervention d) Do not present excess weight as a side effect of a pharmacological treatment that could act as a confounding variable.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from children's weight (z-BMI score) | Change from baseline (pre-intervention) at immediately after 6 months intervention, 12 and 18 months follow-up.
  Rate of overweight and obesity in the children's sample. Instrument: Seca digital (Type 799 and 769) weighing scales.
Change from levels of physical activity | Change from baseline (pre-intervention) at immediately after 6 months intervention and 18 months follow-up.
  Levels of light, moderate and vigorous physical activity. Instrument: accelerometers.
Prevalence of child psychiatric disorders | Baseline (pre-intervention)
  Percent of children with a psychiatric diagnosis according to DSM-5 criteria. Instrument: The Schedule for Affective Disorders and Schizophrenia for School-Age Children Present and Lifetime version.
Change from levels of anxiety symptomatology in children | Change from baseline (pre-intervention) at immediately after 6 months intervention, 12 and 18 months follow-up.
  Questionnaire Spence Children's Anxiety Scale (SCAS): levels of anxiety. Minimum/maximum values: 0-114. Higher scores mean a worse outcome.
Change from levels of depressive symptomatology in children | Change from baseline (pre-intervention) at immediately after 6 months intervention, 12 and 18 months follow-up.
  Questionnaire Children's Depression Inventory (CDI): levels of depressive symptomatology. Minimum/maximum values: 0-54. Spanish risk cut off-point: 19 Higher scores mean a worse outcome.
Change from perceived weight-stigma in children | Change from baseline (pre-intervention) at immediately after 6 months intervention.
  Questionnaire Weight Bias Internalization Scale for Children (WBIS-C). Minimum/maximum score: 11-44 Higher scores on the WBIS-C indicate higher level of weight bias internalization.
Change from incidence of teasing in children | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Perception of Teasing Scale (POTS). It has two factors, weight and competency. Higher scores in each subscale mean a worse outcome (higher prevalence of teasing).
  Perception of Teasing Scale (POTS): Two scales: weight (SUME item1 + item2 + item3 + item4 + item5 + item6) and competency (SUME item7 + item8 + item9 + item10 + item11) Likert Scale 5 points. Maximum score: 30 (weight scale) and 25 (competency scale). Higher scores in each scale mean a worse outcome.
Change from levels of self-esteem in children | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Lawrence's Self-Esteem Questionnaire (LAWSEQ): levels of self-esteem in children. Minimum/maximum value: 0-24. A score below average (score 9) means low self-esteem. A score higher than 9 points means high self-esteem.
Change from emotional regulation in children | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Trait Meta-Mood Scale (TMMS-24). It has three scales: identification, comprehension and regulation of emotions (8 items/scale). Likert Scale 1-5 points. Higher scores in each subscale mean a better outcome.
Change from eating behaviors in children | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Dutch Eating Behaviour Questionnaire for children (DEBQ-C) with scales for restrained, emotional, and external eating. Higher scores in each subscale mean a worse outcome.
Change from levels of perfectionism in children | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Child-Adolescent Perfectionism Scale (CAPS): levels of perfectionism. Subscales of Self-Oriented Perfectionism and Socially Prescribed Perfectionism. The Self-oriented Perfectionism subscale is scored by summing the following items:
  1, 2, 4, 6, 7, 9, 11, 14, 16, 18, 20, 22. The Socially Prescribed Perfectionism subscale is scored by summing the following items: 3, 5, 8, 10, 12, 13, 15, 17, 19, 21. Important: Reverse the following items: 3, 9, 18. Higher scores mean a worse outcome.
Accumulation of psychosocial stress events during childhood | Baseline (pre-intervention)
  Questionnaire: number of psychosocial stress events in school family and social contexts
Change from health habits (nutrition and physical activity) from children and their principal caregiver's | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Semi-structured interview about health habits (nutrition and physical activity)
Change from levels of expressed emotion in family environment | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Family Questionnaire (FQ): incidence of expressed emotion in principal caregiver's (two subscales emotional over-involvement and levels of criticism). Higher scores mean a worse outcome. Risk cut-off point in each subscale: scoring over 23 (criticism) and scoring over 27 (emotional over-involvement).
Change from parental child feeding perceptions, attitudes and practices | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Child Feeding Questionnaire (CFQ): rate of maladaptive parental child feeding perceptions, attitudes and practices. Higher scores mean a worse outcome.
Change from parental educational styles | Change from baseline (pre-intervention) at immediately after intervention, 6, 12 and 18 months follow-up.
  Questionnaire Child's Reports of Parental Behavior Inventory (CRPBI): prevalence and changes of parental educational styles.
  Each parenting style is related to the sum of specific scores on each subscale. Higher scores on each subscale mean a higher prevalence of this educational style.
Change from awareness of the problem and motivation to change about the overweight of their children | Change from baseline (pre-intervention) at immediately after intervention, 6 and 18 months follow-up.
  Questionnaire Change Assessment Scale (URICA): awareness of the problem and motivation to change about the overweight of their children.

SECONDARY OUTCOMES:
Primary Caregiver's Body Mass Index (BMI) | Change from baseline (pre-intervention) at immediately after intervention, 12 and 18 months follow-up.
  Body Mass Index (weight/height)
Family socio-demographic variables | Baseline (pre-intervention)
  Semi-structured interview: parents' age, marital status, nationality educational level, current job, socioeconomic status.
Health habits and eating patterns in principal caregivers. | Baseline (pre-intervention)
  Semi-structure interview carried out with principal caregivers to explore their feeding routine and the presence/absence of eating disorders symptomatology
Change of eating behaviors in adults | Change from baseline (pre-intervention) at immediately after intervention, 6 and 18 months follow-up.
  Dutch Eating Behaviour Questionnaire (DEBQ) with scales for restrained, emotional, and external eating. Higher scores in each subscale mean a worse outcome.
Levels of psychological well-being in principal caregivers | Baseline (pre-intervention)
  Questionnaire: Stressful Life Events and Daily Hassles (SRRS). A total value for stressful life events can be worked out by adding up the scores for each event experienced over a 12 month period. If a person has less the 150 life change units they have a 30% chance of suffering from stress. 150 - 299 life change units equates to a 50% chance of suffering from stress. Over 300 life units means a person has an 80% chance of developing a stress related illness.
Levels of psychological well-being in principal caregivers | Change from baseline (pre-intervention) at immediately after intervention, 6 and 18 months follow-up.
  Levels of depressive symptomatology. Beck's Depression Inventory (BDI). Higher scores mean a worse outcome.
Child executive functions screening | Baseline (pre-intervention)
  Questionnaire Behavior Rating Inventory of Executive Function (BRIEF2-F): screening of executive functioning in children. This questionnaire is answered by principal caregiver's. Eight clinical scales (Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor) and an overall score. All 63 items are rated in terms of frequency on a 3-point scale: 0 (never), 1 (sometimes), 2 (often).

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Sepúlveda, PhD, Principal Investigator — Universidad Autonoma de Madrid
Locations (1):
- Ms. Sepúlveda. Coordinator of ENTREN Program. ANOBAS Group Research. School of Psychology (AUM) Web: www.anobas.es Contact: anarosa.sepulveda@uam.es/programaentren@gmail.com, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study protocol is available. The structure of the program and the specific content of the sessions will be available in a published guidebook. Upon prior request, a document with the interpretation of the items in Statistical Package for the Social Sciences (SPSS) databases, a description of the instruments and outcomes variables included in this study, may also be provided. PhD. Ana Rosa Sepúlveda will be the responsible of reviewing all request, and taking a final decision. Criteria for reviewing requests: National and international Research Groups related to childhood obesity or eating disorders. Types of analyses: replica of ENTREN's Randomised controlled trials (RCT) in other countries or meta-analyses studies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will become available from December of 2021. Period of availability: unlimited after publication. Request and a revision of the request are both necessary conditions.
Access Criteria: The study protocol will also be available. The structure of the program and the specific content of the sessions will be available in a published guidebook. Upon prior request, a document with the interpretation of the items in SPSS databases, a description of the instruments and outcomes variables included in this study, may also be provided. PhD. Ana Rosa Sepúlveda will be the responsible of reviewing all request, and taking a final decision. Criteria for reviewing requests: National and international Research Groups related to childhood obesity or eating disorders. Types of analyses: replica of ENTREN's RCT in other countries or meta-analyses studies.

REFERENCES:
- [Background] Sepulveda AR, Solano S, Blanco M, Lacruz T, Graell M. Prevalence of childhood mental disorders in overweight and obese Spanish children: Identifying loss of control eating. Psychiatry Res. 2018 Sep;267:175-181. doi: 10.1016/j.psychres.2018.06.019. Epub 2018 Jun 8. PMID 29909128
- [Background] Blanco M, Sepulveda AR, Lacruz T, Parks M, Real B, Martin-Peinador Y, Roman FJ. Examining Maternal Psychopathology, Family Functioning and Coping Skills in Childhood Obesity: A Case-Control Study. Eur Eat Disord Rev. 2017 Sep;25(5):359-365. doi: 10.1002/erv.2527. Epub 2017 Jun 1. PMID 28568706
- [Background] Blanco M, Veiga OL, Sepulveda AR, Izquierdo-Gomez R, Roman FJ, Lopez S, Rojo M. [Family environment, physical activity and sedentarism in preadolescents with childhood obesity: ANOBAS case-control study]. Aten Primaria. 2020 Apr;52(4):250-257. doi: 10.1016/j.aprim.2018.05.013. Epub 2019 Mar 18. Spanish. PMID 30898477
- [Background] Hemmingsson E. A new model of the role of psychological and emotional distress in promoting obesity: conceptual review with implications for treatment and prevention. Obes Rev. 2014 Sep;15(9):769-79. doi: 10.1111/obr.12197. Epub 2014 Jun 16. PMID 24931366
- [Background] Robertson W, Fleming J, Kamal A, Hamborg T, Khan KA, Griffiths F, Stewart-Brown S, Stallard N, Petrou S, Simkiss D, Harrison E, Kim SW, Thorogood M. Randomised controlled trial evaluating the effectiveness and cost-effectiveness of 'Families for Health', a family-based childhood obesity treatment intervention delivered in a community setting for ages 6 to 11 years. Health Technol Assess. 2017 Jan;21(1):1-180. doi: 10.3310/hta21010. PMID 28059054
- [Result] Sepulveda AR, Solano S, Blanco M, Lacruz T, Veiga O. Feasibility, acceptability, and effectiveness of a multidisciplinary intervention in childhood obesity from primary care: Nutrition, physical activity, emotional regulation, and family. Eur Eat Disord Rev. 2020 Mar;28(2):184-198. doi: 10.1002/erv.2702. Epub 2019 Dec 4. PMID 31802570
- [Result] Rojo M, Lacruz T, Solano S, Vivar M, Del Rio A, Martinez J, Foguet S, Marin M, Moreno-Encinas A, Veiga OL, Cabanas V, Rey C, Graell M, Sepulveda AR. ENTREN-F family-system based intervention for managing childhood obesity: Study protocol for a randomized controlled trial at primary care. Obes Res Clin Pract. 2022 Jul-Aug;16(4):319-329. doi: 10.1016/j.orcp.2022.07.001. Epub 2022 Jul 22. PMID 35871907
- [Result] Rojo M, Lacruz T, Solano S, Gutierrez A, Beltran-Garrayo L, Veiga OL, Graell M, Sepulveda AR. Family-reported barriers and predictors of short-term attendance in a multidisciplinary intervention for managing childhood obesity: A psycho-family-system based randomised controlled trial (ENTREN-F). Eur Eat Disord Rev. 2022 Nov;30(6):746-759. doi: 10.1002/erv.2913. Epub 2022 May 28. PMID 35644038
- See also: Research Group webpage. ANOBAS Research Team website (Faculty of Psychology - AUM). Three lines of research currently active (EDs, childhood obesity and body dysmorphia). Information about team members, the ENTREN program and resources for professionals. — http://www.anobas.es

DOCUMENTS (3):
  • Study Protocol (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT04465799/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT04465799/SAP_001.pdf
  • Informed Consent Form (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/99/NCT04465799/ICF_002.pdf